CLINICAL TRIAL: NCT07373782
Title: Reducing Cardiac Radiation Dose in Continuous Positive Airway Pressure (CPAP) Assisted Radiotherapy in Breast Cancer: a Prospective Non-Randomized Clinical Trial
Brief Title: Continuous Positive Airway Pressure (CPAP) Assisted Radiotherapy in Breast Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: VitalAire (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: S68702
Record Dates: First submitted 2025-12-10; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3)
Keywords: breast cancer; radiotherapy; cpap; continuous positive airway pressure; dosimetry; toxicity
MeSH Terms: conditions — Breast Neoplasms; Microcephaly, Primary Autosomal Recessive, 6 | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: prospective clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CPAP-addition (Experimental): CPAP is added to standard of care
  Interventions: Device: Continuous Positive Airway Pressure (CPAP)
- Standard of care (No Intervention): Right sided or 70 years or older: Free Breathing Left sided and younger than 70 years old: Deep Inspiration Breath Hold

INTERVENTIONS:
Device: Continuous Positive Airway Pressure (CPAP) — Positive airway pressure (15cmH2O) delivered by a CPAP-device
  Arms: CPAP-addition

SUMMARY:
This study is a prospective, non-randomized clinical study aimed at investigating the potential benefits of continuous positive airway pressure (CPAP) support during radiotherapy for breast cancer. CPAP is a device commonly used to support breathing, for example in patients with sleep apnea. The investigators expect a reduction in radiation doses to the heart and/or lungs with CPAP-supported radiotherapy compared to standard radiotherapy (without CPAP), which may also lead to a decrease in radiation-induced heart and/or lung conditions in the long term. The study will also examine how the use of a CPAP device can be implemented in daily radiotherapy practice.

DETAILED DESCRIPTION:
Patients undergoing breast conserving surgery for invasive or in situ BC and requiring adjuvant RT are prospectively enrolled -either left-sided cases with or without regional nodal irradiation (RNI), or right-sided cases requiring RNI. Each patient undergoes an additional CT simulation with continuous positive airway pressure (CPAP) (15cm H20) -in free breathing (FB) for right-sided cases and in deep inspiration breath hold (DIBH) for left-sided cases. Left-sided patients unable to perform DIBH are evaluated in FB. Two RT plans (with and without CPAP) are dosimetrically compared. If CPAP reduces mean heart or CLB dose by ≥0.5 Gy, or mean lung dose by ≥1 Gy, treatment is delivered with CPAP. Patient comfort is assessed through surveys.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
2. At least 40 years of age and 80 years or younger at the time of signing the Informed Consent Form (ICF)
3. Female patients
4. Patients that underwent breast conserving surgery (BCS)
5. Left-sided invasive BC / in situ carcinoma with indication for adjuvant RT (<70 years old)
6. Left-sided invasive BC with indication for adjuvant locoregional RT (including RT of the regional lymph nodes) (70-80 years old)
7. Right-sided invasive BC with indication for adjuvant locoregional RT (including RT of the regional lymph nodes)
8. Prior chemotherapy allowed
9. Prior immunotherapy allowed
10. Prior / concomitant hormonal therapy allowed
11. Prior / concomitant HER2-targeted therapy allowed

Exclusion Criteria:

1. Patient has active bullous lung disease, bypassed upper airway, pneumothorax, cerebral spinal fluid leaks, abnormalities of the cribriform plate (contra-indications for the use of CPAP)
2. Patient has history of major head trauma and/or pneumocephalus (contra-indications for the use of CPAP)
3. Any disorder, which in the investigator's opinion might jeopardise participant's safety or compliance with the CIP.
4. Female who is pregnant, breast-feeding or intends to become pregnant (which is a contra-indication for RT in general)
5. Male BC patients
6. Patients that underwent mastectomy Patients whose initial tumor was located just beneath the skin (defined as being less than 28mm below the breast surface), indicating the need for an electron boost
7. Patients requiring RT boost on positive lymph nodes
8. Distant metastasis
9. Breast implants in situ
10. Right-sided in situ carcinoma
11. Right-sided invasive BC only requiring local adjuvant RT (without irradiation of the regional lymph nodes, because the presumed benefit on cardiac doses of local right-sided breast irradiation is assumed to be rather small because of the left anatomical position of the heart)
12. Bilateral BC
13. Concomitant use of chemotherapy during RT
14. Substantial comorbidities, incompatible with RT or CPAP use, estimated by the treating radiation oncologist
15. Insufficient arm mobility to perform comfortable arm positioning in radiation treatment position, evaluated by the treating radiation oncologist
16. Other active oncological disease / treatment with the exception of non-melanoma skin cancer
17. Previous RT with overlapping RT fields with actual target volume

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Mean heart dose | From enrollment to the end of treatment at +/-8 weeks
  Potential change of mean radiation dose to the heart

SECONDARY OUTCOMES:
Doses to cardiac substructures | From enrollment to the end of treatment at +/-8 weeks
  Potential change in radiation dose to cardiac substructures
Mean lung dose | From enrollment to the end of treatment at +/-8 weeks
  Potential change in mean radiation dose to the lungs
Mean contralateral breast dose | From enrollment to the end of treatment at +/-8 weeks
  Potential change in mean radiation dose to the contralateral breast
Liver dose | From enrollment to the end of treatment at +/-8 weeks
  Potential change in radiation dose to the liver
Patient comfort | From enrollment to the end of treatment at +/-8 weeks
  Patient comfort assessed through patient questionnaires (Likert scale: Strongly disagree - disagree - neutral - agree - strongly agree)
Reproducibility and accuracy of CPAP-assisted radiotherapy | From enrollment to the end of treatment at +/-8 weeks
  Compare reproducibility and accuracy between standard and CPAP-assisted RT by using surface scanning and daily cone beam CT (CBCT) parameters
DIBH performance | From enrollment to the end of treatment at +/-8 weeks
  To compare DIBH performance between standard and CPAP-assisted RT for left-sided BC by using surface scanning and daily CBCT parameters
Time-effectiveness | From enrollment to the end of treatment at +/-8 weeks
  To compare time-effectiveness between standard and CPAP-assisted RT
  * Set-up time
  * Matching time
  * Radiation time

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT07373782/Prot_SAP_000.pdf